CLINICAL TRIAL: NCT05918445
Title: Phase Ib/IIa Safety and Efficacy of PM8002, a Bispecific Antibody Targeting PD-L1 and VEGF-A, as a Monotherapy in Patients With Advanced Solid Tumors
Brief Title: PM8002 in the Treatment of Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biotheus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PM8002-A001
Record Dates: First submitted 2023-05-30; First posted 2023-06-26 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PM8002 (Experimental): PM8002 IV every 2 weeks(q2w) or every 3 weeks(q3w)
  Interventions: Drug: PM8002

INTERVENTIONS:
Drug: PM8002 — IV infusion

SUMMARY:
This study is to characterize the safety, tolerability, pharmacokinetics (PK), immunogenicity, pharmacodynamics (PD) and anti-tumor activity of PM8002, a PD-L1/VEGF bispecific antibody, as a single agent in adult subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in clinical study; fully understand the study and sign informed consent voluntarily; willing to follow and able to complete all test procedures;
2. Male or female aged 18 to 75 years;
3. Patients with malignant tumor confirmed by histology or cytology;
4. The toxicity of previous anti-tumor therapy has not been alleviated；
5. Adequate organ function；
6. ECOG score was 0-1;
7. Expected survival >=12 weeks;
8. According to RECIST 1.1 criteria, at least 1 measurable lesion that has not been previously treated locally.

Exclusion Criteria:

1. History of severe allergic disease, severe allergy to drugs or known allergy to any component of the drug in this study;
2. Evidence of major coagulopathy or other obvious risk of bleeding;
3. Patients are experiencing a clear interstitial lung disease or non-infectious pneumonia, unless it is caused by local radiotherapy;
4. Patients with uncontrolled brain metastases should be excluded from this clinical trial;
5. Patients ever experienced other active malignant tumors within 5 years prior to the study treatment;
6. Prior allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
7. Known history of alcohol abuse, psychotropic drug abuse or drug abuse;
8. Syphilis antibody positive;
9. Patients with active tuberculosis (TB) are excluded;
10. Pregnant or lactating women;
11. Other conditions lead to inappropriate to participate in this study as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with DLTs | During the first three weeks of treatment with PM8002
  DLTs will be assessed during the dose-escalation phase and are defined as toxicities that meet pre-defined severity criteria and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, intercurrent illness, or concomitant medications that occurs within the first cycle (3weeks) of treatment.
Treatment related adverse events (TRAEs) | Up to 30 days after last treatment
  The incidence and severity of TRAEs graded according to NCI-CTCAE v5.0
Objective response rate (ORR) | Up to approximately 2 years
  Objective response rate (ORR) is the proportion of subjects with complete response (CR) or partial response (PR), based on RECIST v1.1.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to approximately 2 years
  DCR is defined as the proportion of subjects with CR, PR, or stable disease(SD) based on RECIST v1.1.
Duration of response (DoR) | Up to approximately 2 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression (based on RECIST v1.1). for subjects with no documented disease progression, the deadline is the data of the last examination.
Overall survival (OS) | Up to approximately 2 years
  OS is the time from the date of first dosing date to death due to any cause.
Progression-free survival (PFS) | Up to approximately 2 years
  Progression-free survival is defined as the time from the start of treatment with PM8002 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Anti-drug antibody (ADA) | Up to 30 days after last treatment
  To evaluate the incidence of ADA to PM8002.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, Principal Investigator — Shanghai Orient Hospital
Locations (39):
- China (39):
  - Baoji Central Hospital, Baoji
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Peking University Cancer Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - The First Hospital of Jilin University, Changchun
  - Changde First People's Hospital, Changde
  - Hunan Provincial People's Hospital, Changsha
  - The First People's Hospital of Changzhou, Changzhou
  - Chengdu Integrated TCM& Western Medicine Hospital, Chengdu
  - Sichuan Cancer Hospital, Chengdu
  - Chongqing Cancer Hospital, Chongqing
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - The Southwest Hospital of AMU, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Provincial Hospital, Hefei
  - Linyi Cancer Hospital, Linyi
  - Jiangsu Province Hospital, Nanjing
  - Shanghai Orient Hospital, Shanghai
  - Shanghai Sixth People's Hospital, Shanghai
  - Shengjing Hospital of China Medical University, Shengjing
  - Liaoning Cancer Hospital, Shenyang
  - The First Hospital of China Medical University, Shenyang
  - The People's Hospital of Liaoning Province, Shenyang
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang
  - Shanxi Bethune Hospital, Taiyuan
  - Shanxi Provincial Cancer Hospital, Taiyuan
  - Taizhou Hospital of Zhejiang Province, Taizhou
  - The Second Hospital of Tianjin Medical University, Tianjin
  - Hubei Cancer Hospital, Wuhan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Xi 'an International Medical Center Hospital, Xi'an
  - Yantai Yuhuangding Hospital, Yantai
  - Yibin Second People's Hospital, Yibin
  - Henan Cancer Hospital, Zhengzhou
  - The first affilated hospital of zhengzhou university, Zhengzhou
  - Zhujiang Hospital of Southern Medical University, Zhujiang

IPD SHARING:
Plan to Share IPD: Yes
The data will be published or presented for publications (poster, abstract, articles or papers) or any presentations.
Time Frame: After the trial completed
Access Criteria: NCI is committed to sharing data in accordance with NIH policy.